CLINICAL TRIAL: NCT02882711
Title: A Naturalistic Study of Serial Infusion of Low-dose Ketamine for Treatment Resistant Depressive Disorders in an Academic Psychiatric Hospital: The UTHealth Ketamine Project
Brief Title: The UTHealth Ketamine Project
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Increasing off-label practice of IV ketamine administration for treatment-resistant depression.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Salih Selek, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0020
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder | interventions — Ketamine

ARMS (1):
- ketamine (Experimental)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine will be infused (slow IV infusions of ketamine (0.5 mg/kg) over 40 minutes) twice weekly over a period of 4 weeks and weekly for the following 4 weeks of the study treatment period (8 weeks total).

SUMMARY:
The primary objective of this study is to determine the effectiveness of serial infusions of intravenous (IV) ketamine in adults with treatment resistant depression (TRD).

DETAILED DESCRIPTION:
Thus, in the current study we want to naturalistically explore the antidepressant effects of serial slow IV infusions (40 minutes) of ketamine at a dose of 0.5 mg/kg, over a treatment period of 8 weeks in an academic psychiatric hospital. This is a minimal sedation treatment. The primary outcome measure of this study will be remission estimated based on the severity of depressive scores. After the 8 weeks of treatment, there will be a four week observational period. During the observational period, participants will receive treatment as usual and will be contacted over the phone for follow-up questions regarding their overall health status, mood and clinical state. They will also complete a neurocognitive task at the end of the 4 week observational period

ELIGIBILITY:
Inclusion Criteria:

* patients with major depressive disorder (MDD) or bipolar disorder (BD)
* patients with documented treatment resistant disorder (TRD) (according to Diagnostic Statistical Manual (DSM-IV TR)), and who have failed (defined as patient does not reach remission within the 8 week trial of an antidepressant or combination at a therapeutic dose) of at least two trials of first line evidence-based treatments and/or electroconvulsive therapy (ECT)

Exclusion Criteria:

* Being younger than 18 of age or older than 65.
* Diagnosed with intellectual disability, e.g. mental retardation (MR), neurodegenerative diseases, e.g. early-onset neurocognitive disturbances such as frontotemporal dementia (FTD) or behavioral disorders, e.g. adult onset Attention Deficit Hyperactivity Disorder (ADHD).
* Diagnosed with bipolar disorder not otherwise specified (BD-NOS) or rapid cycling BD
* Diagnosed with personality disorders (PD).
* Previously or currently diagnosed with psychosis (schizoaffective disorder - SAD) or schizophrenia - SCZ).
* Current major medical problems that affect brain anatomy, neurochemistry, or function, e.g., obstructive sleep apnea requiring Continuous Positive Airway Pressure (CPAP), liver insufficiency, kidney insufficiency, cardiovascular problems, systemic infections, cancer, auto-immune diseases, and any brain disorder (seizure disorder, stroke, dementia, degenerative neurologic diseases); history of any brain diseases, including seizures, stroke, meningitis, encephalitis, dementia, degenerative brain diseases, and head injury with loss of consciousness for any period of time.
* Diagnosed specifically with a cardiovascular disorders such as Arrhythmias, Chronic Heart Failure, Myocardial Infarction (MI) or suffering from Chronic Obstructive Pulmonary Disease (COPD) or asthma. Suffering from uncontrolled hypertension or diastolic BP over 100. Cardiac clearance prior to enrolling in the study/medical records from physician will be required per patient's primary care physician (PCP).
* Patients with increased risk of laryngospasm, active upper respiratory infections, respiratory depression, increased intracranial pressure, hyperthyroidism, or porphyria.
* Current substance abuse or dependence. Only patients who achieved stable, full remission for at least 6 months will be included.
* Pregnancy or Breast feeding. All female in reproductive age will undergo pregnancy tests. Female participants will be required to provide evidence of use of contraceptives during the course of the study.
* Unable to understand the design and requirements of the study
* Unable to sign the informed consent for any reason
* An assigned responsible adult has provided assent to assist in patient's study participation. The responsible adult agrees to be present at each study appointment as well as provide transportation to study appointments for the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salih Selek, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants who were enrolled met exclusion criteria and therefore did not start the study.
Period: Overall Study
Arm/Group | Ketamine
Started | 6
Completed | 2
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Safety Will be Measured Through Number of Adverse Events
Time Frame: Baseline through week 12
Population: This data was only collected for the 2 participants who completed the study.
Measure: Number; unit: adverse events
Arm/Group | Ketamine
Number analyzed (Participants) | 2
adverse events | 2

2. Secondary Outcome: Efficacy of Treatment Will be Measured on of Clinical Global Impressions (CGI)
Time Frame: Baseline, week 8, week 12
Population: Clinical Global Impressions (CGI) scale data was not collected for any participant
Arm/Group | Ketamine
Number analyzed (Participants) | 0

3. Secondary Outcome: Severity of Depressive Symptoms as Assessed by the PHQ-9
Description: The Patient Health Questionnaire (PHQ)-9 is the 9-item depression module from the full Patient Health Questionnaire (PHQ) PHQ-9 total score ranges from 0 to 27 (each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day)), and a higher score indicates greater depression.
Time Frame: Baseline, week 8, week 12
Population: PHQ-9 data was collected at baseline for all 6 participants who started the study. PHQ-9 data was not collected at week 8 or week 12 for 4 participants, per study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 6
units on a scale
  Baseline | 12.67 (9.501)
  Week 8: number analyzed (Participants) | 2
  Week 8 | 5 (5.657)
  Week 12: number analyzed (Participants) | 2
  Week 12 | 5 (5.657)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=6)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=6)
dissociation (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Not reaching the target number of participants needed to achieve target power

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02882711/Prot_SAP_000.pdf